CLINICAL TRIAL: NCT00005502
Title: Coronary Disease Morbidity and Mortality in a Population
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Veronique L. Roger, Consultant- Cardiology NonInvasive, Mayo Clinic
Other Study IDs: 632-01; R01HL059205 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, serum and white blood cells are stored for future research projects
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Residents of Olmsted County, MN with elevated Troponins: Anyone admitted to St Marys or Rochester Methodist Hospitals who have an elevated troponin during their hospitalization and are residents of Olmsted County, MN

SUMMARY:
To study the entire population of Olmsted County, Minnesota, including all age categories, to examine the secular trends in coronary heart disease (CHD) mortality, myocardial infarction (MI) incidence, and natural history, including MI severity, case fatality and post-MI morbidity. Also, to examine the time trends in the prevalence of CHD at post-mortem because of the uniquely high autopsy rate in Olmsted County.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease remains the leading cause of death in the U.S. Despite an encouraging decline in age-adjusted coronary heart disease (CHD) mortality, prevalent CHD continues to represent a major health burden, particularly in the elderly population. Most community surveillance programs, however, cannot fully characterize this problem because they are restricted to an upper age limit of 74 years and thus do not include the events occurring in an increasingly growing part of the population. Observational studies have questioned the existence of a change over time in the prevalence of anatomic coronary disease either at post-mortem examination or at coronary angiography. This remains to be further examined in a population-based setting. In addition, the natural history of myocardial infarction (MI) in the reperfusion area is unknown; in particular, there are no population-based data on the incidence of post-MI heart failure.

DESIGN NARRATIVE:

The records of all Olmsted County residents with a hospital discharge diagnosis of MI between 1979 and 1999 were reviewed, and standard epidemiologic MI validation criteria were applied; post-MI outcome over time was determined, including post-MI heart failure, angina, 30 day case fatality and long-term survival. In parallel with the analysis of time trends in CHD mortality, the autopsy reports were reviewed to examine whether the prevalence of coronary disease at autopsy has changed over time. These studies provided an assessment of the clinical and anatomical manifestations of CHD, including the outcome of acute MI, over a time period characterized by intensified primary prevention efforts and major changes in the treatment of acute CHD.

The study was renewed in July 2002 to continue surveillance of acute coronary heart disease events in order to address issues surrounding the diagnostic precision and risk stratification potential of troponin and high sensitivity C reactive protein (CRP) and to monitor secular trends in severity and treatment modalities. Novel approaches to the procurement of carefully timed blood samples allow direct measurement of the increase in number of cases of myocardial infarction using the new biomarker, troponin. An examination will be made of the prognostic value of quantitative peak troponin measured at 24 to 36 hours and high sensitivity C reactive protein measured early after symptom onset in the myocardial infarction cohort.

ELIGIBILITY:
All residents of Olmsted County, MN who are hospitalized and have an elevated Troponin level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All residents of Olmsted County, MN who are hospitalized and have an elevated Troponin level.Non-residenst of Olmsted County are excluded.
Sampling Method: Probability Sample
Enrollment: 5476 (Actual)
Dates: Start 2002-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To measure the number of Olmsted County,MN residents who have a Myocardial Infarction and Unstable Angina. | 1979 through 2012

SECONDARY OUTCOMES:
To measure the survival of Olmsted County, MN residents after having a Myocardial Infarction or Unstable Angina event | 1979-2012

OTHER OUTCOMES:
To examine the value of biomarkers on prediction of risks in Olmsted County, MN residents who have a Myocardial Infarction or Unstable Angina | 2002-2012

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Roger, Principal Investigator — Mayo Foundation
Locations (2):
- United States (2):
  - St Marys Hospital, Rochester, Minnesota
  - Rochester Methodist Hospital, Rochester, Minnesota

REFERENCES:
- [Background] Roger VL, Farkouh ME, Weston SA, Reeder GS, Jacobsen SJ, Zinsmeister AR, Yawn BP, Kopecky SL, Gabriel SE. Sex differences in evaluation and outcome of unstable angina. JAMA. 2000 Feb 2;283(5):646-52. doi: 10.1001/jama.283.5.646. PMID 10665705
- [Background] Roger VL, Jacobsen SJ, Weston SA, Bailey KR, Kottke TE, Frye RL. Trends in heart disease deaths in Olmsted County, Minnesota, 1979-1994. Mayo Clin Proc. 1999 Jul;74(7):651-7. doi: 10.4065/74.7.651. PMID 10405692
- [Background] Roger VL, Weston SA, Killian JM, Pfeifer EA, Belau PG, Kottke TE, Frye RL, Bailey KR, Jacobsen SJ. Time trends in the prevalence of atherosclerosis: a population-based autopsy study. Am J Med. 2001 Mar;110(4):267-73. doi: 10.1016/s0002-9343(00)00709-9. PMID 11239844
- [Background] Goraya TY, Jacobsen SJ, Belau PG, Weston SA, Kottke TE, Roger VL. Validation of death certificate diagnosis of out-of-hospital coronary heart disease deaths in Olmsted County, Minnesota. Mayo Clin Proc. 2000 Jul;75(7):681-7. doi: 10.4065/75.7.681. PMID 10907382
- [Background] Targonski P, Jacobsen SJ, Weston SA, Leibson CL, Pfeifer E, Nemetz P, Roger VL. Referral to autopsy: effect of antemortem cardiovascular disease: a population-based study in Olmsted County, Minnesota. Ann Epidemiol. 2001 May;11(4):264-70. doi: 10.1016/s1047-2797(00)00220-9. PMID 11306345
- [Background] Hellermann JP, Reeder GS, Jacobsen SJ, Weston SA, Killian JM, Roger VL. Longitudinal trends in the severity of acute myocardial infarction: a population study in Olmsted County, Minnesota. Am J Epidemiol. 2002 Aug 1;156(3):246-53. doi: 10.1093/aje/kwf034. PMID 12142259
- [Background] Roger VL, Killian J, Henkel M, Weston SA, Goraya TY, Yawn BP, Kottke TE, Frye RL, Jacobsen SJ. Coronary disease surveillance in Olmsted County objectives and methodology. J Clin Epidemiol. 2002 Jun;55(6):593-601. doi: 10.1016/s0895-4356(02)00390-6. PMID 12063101
- [Background] Roger VL, Jacobsen SJ, Weston SA, Goraya TY, Killian J, Reeder GS, Kottke TE, Yawn BP, Frye RL. Trends in the incidence and survival of patients with hospitalized myocardial infarction, Olmsted County, Minnesota, 1979 to 1994. Ann Intern Med. 2002 Mar 5;136(5):341-8. doi: 10.7326/0003-4819-136-5-200203050-00005. PMID 11874305
- [Background] Goraya TY, Leibson CL, Palumbo PJ, Weston SA, Killian JM, Pfeifer EA, Jacobsen SJ, Frye RL, Roger VL. Coronary atherosclerosis in diabetes mellitus: a population-based autopsy study. J Am Coll Cardiol. 2002 Sep 4;40(5):946-53. doi: 10.1016/s0735-1097(02)02065-x. PMID 12225721
- [Background] Goraya TY, Jacobsen SJ, Kottke TE, Frye RL, Weston SA, Roger VL. Coronary heart disease death and sudden cardiac death: a 20-year population-based study. Am J Epidemiol. 2003 May 1;157(9):763-70. doi: 10.1093/aje/kwg057. PMID 12727669
- [Background] Hellermann JP, Goraya TY, Jacobsen SJ, Weston SA, Reeder GS, Gersh BJ, Redfield MM, Rodeheffer RJ, Yawn BP, Roger VL. Incidence of heart failure after myocardial infarction: is it changing over time? Am J Epidemiol. 2003 Jun 15;157(12):1101-7. doi: 10.1093/aje/kwg078. PMID 12796046
- [Background] Hellermann JP, Jacobsen SJ, Reeder GS, Lopez-Jimenez F, Weston SA, Roger VL. Heart failure after myocardial infarction: prevalence of preserved left ventricular systolic function in the community. Am Heart J. 2003 Apr;145(4):742-8. doi: 10.1067/mhj.2003.187. PMID 12679774
- [Background] Singh M, Reeder GS, Jacobsen SJ, Weston S, Killian J, Roger VL. Scores for post-myocardial infarction risk stratification in the community. Circulation. 2002 Oct 29;106(18):2309-14. doi: 10.1161/01.cir.0000036598.12888.de. PMID 12403659
- [Background] Hellermann JP, Jacobsen SJ, Gersh BJ, Rodeheffer RJ, Reeder GS, Roger VL. Heart failure after myocardial infarction: a review. Am J Med. 2002 Sep;113(4):324-30. doi: 10.1016/s0002-9343(02)01185-3. PMID 12361819
- [Background] Roger VL, Jacobsen SJ, Weston SA, Pellikka PA, Miller TD, Bailey KR, Gersh BJ. Sex differences in evaluation and outcome after stress testing. Mayo Clin Proc. 2002 Jul;77(7):638-45. doi: 10.4065/77.7.638. PMID 12108601
- [Background] Jokhadar M, Jacobsen SJ, Reeder GS, Weston SA, Roger VL. Sudden death and recurrent ischemic events after myocardial infarction in the community. Am J Epidemiol. 2004 Jun 1;159(11):1040-6. doi: 10.1093/aje/kwh147. PMID 15155288
- [Background] Lopez-Jimenez F, Jacobsen SJ, Reeder GS, Weston SA, Meverden RA, Roger VL. Prevalence and secular trends of excess body weight and impact on outcomes after myocardial infarction in the community. Chest. 2004 Apr;125(4):1205-12. doi: 10.1378/chest.125.4.1205. PMID 15078726
- [Background] Lopez-Jimenez F, Goraya TY, Hellermann JP, Jacobsen SJ, Reeder GS, Weston SA, Roger VL. Measurement of ejection fraction after myocardial infarction in the population. Chest. 2004 Feb;125(2):397-403. doi: 10.1378/chest.125.2.397. PMID 14769715
- [Background] Witt BJ, Jacobsen SJ, Weston SA, Killian JM, Meverden RA, Allison TG, Reeder GS, Roger VL. Cardiac rehabilitation after myocardial infarction in the community. J Am Coll Cardiol. 2004 Sep 1;44(5):988-96. doi: 10.1016/j.jacc.2004.05.062. PMID 15337208
- [Background] Perschbacher JM, Reeder GS, Jacobsen SJ, Weston SA, Killian JM, Slobodova A, Roger VL. Evidence-based therapies for myocardial infarction: secular trends and determinants of practice in the community. Mayo Clin Proc. 2004 Aug;79(8):983-91. doi: 10.4065/79.8.983. PMID 15301324
- [Background] Bursi F, Enriquez-Sarano M, Nkomo VT, Jacobsen SJ, Weston SA, Meverden RA, Roger VL. Heart failure and death after myocardial infarction in the community: the emerging role of mitral regurgitation. Circulation. 2005 Jan 25;111(3):295-301. doi: 10.1161/01.CIR.0000151097.30779.04. Epub 2005 Jan 17. PMID 15655133
- [Background] Hellermann JP, Jacobsen SJ, Redfield MM, Reeder GS, Weston SA, Roger VL. Heart failure after myocardial infarction: clinical presentation and survival. Eur J Heart Fail. 2005 Jan;7(1):119-25. doi: 10.1016/j.ejheart.2004.04.011. PMID 15642543
- [Background] Witt BJ, Brown RD Jr, Jacobsen SJ, Weston SA, Yawn BP, Roger VL. A community-based study of stroke incidence after myocardial infarction. Ann Intern Med. 2005 Dec 6;143(11):785-92. doi: 10.7326/0003-4819-143-11-200512060-00006. PMID 16330789
- [Background] Leibson CL, Burke JP, Ransom JE, Forsgren J, Melton J 3rd, Bailey KR, Palumbo PJ. Relative risk of mortality associated with diabetes as a function of birth weight. Diabetes Care. 2005 Dec;28(12):2839-43. doi: 10.2337/diacare.28.12.2839. PMID 16306542
- [Background] Miller TD, Roger VL, Hodge DO, Gibbons RJ. A simple clinical score accurately predicts outcome in a community-based population undergoing stress testing. Am J Med. 2005 Aug;118(8):866-72. doi: 10.1016/j.amjmed.2005.03.013. PMID 16084179
- [Background] Tleyjeh IM, Steckelberg JM, Murad HS, Anavekar NS, Ghomrawi HM, Mirzoyev Z, Moustafa SE, Hoskin TL, Mandrekar JN, Wilson WR, Baddour LM. Temporal trends in infective endocarditis: a population-based study in Olmsted County, Minnesota. JAMA. 2005 Jun 22;293(24):3022-8. doi: 10.1001/jama.293.24.3022. PMID 15972564
- [Background] Bursi F, Rocca WA, Killian JM, Weston SA, Knopman DS, Jacobsen SJ, Roger VL. Heart disease and dementia: a population-based study. Am J Epidemiol. 2006 Jan 15;163(2):135-41. doi: 10.1093/aje/kwj025. Epub 2005 Nov 17. PMID 16293716